CLINICAL TRIAL: NCT02656056
Title: Assessing the Role of a Fermented Soy Extract in Inflammation and the Human Microbiome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: BESO Biological Research, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1507016139
Record Dates: First submitted 2016-01-06; First posted 2016-01-14 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Food

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lean Adults (Experimental): Adults with a BMI between 21-25 will consume 8 oz of the fermented soybean beverage, twice daily.
  Interventions: Other: Food: (Q-Can Plus fermented soybean beverage)
- Obese Adults (Experimental): Adults with a BMI between 32-37 will consume 8 oz of the fermented soybean beverage, twice daily.
  Interventions: Other: Food: (Q-Can Plus fermented soybean beverage)

INTERVENTIONS:
Other: Food: (Q-Can Plus fermented soybean beverage) — Fermented soybean beverage. Dose is 8 oz, twice daily.

SUMMARY:
The consumption of fermented soy foods can alter the human microbiome and may confer health benefits. Researchers propose a line of inquiry to assess the effects of Q-Can Plus ("QC") fermented soy beverage in humans, assessing immunological, microbiological, and clinical parameters.

DETAILED DESCRIPTION:
The study will start with a detailed testing of the microorganisms present in the QC fermented soy liquid, using deep sequencing. Subsequently, the researchers will determine the effect of the QC fermented soy product on the microbiome and inflammation in lean and obese individuals, as obese individuals are known to have dysbiosis. The work on inflammatory changes will be supplemented by studies to investigate the cellular and molecular mechanistic pathways responsible for the biological action of QC fermented soy liquid.

ELIGIBILITY:
Inclusion Criteria:

* Adults (aged between 18 and 70) that are obese (BMI 32-37) (n=10)
* Adults (aged between 18 and 70) that are lean (BMI 21-25) (n=10)

Exclusion Criteria:

* Allergy to soy or soy derivatives.
* Patients will be excluded if they had abdominal surgeries (excluding cholecystectomy, appendectomy, hysterectomy, and hernia repair).
* History of inflammatory bowel disease (e.g., ulcerative colitis, Crohn's disease) and/or gastrointestinal bleeding.
* Medications: Antibiotics, probiotics, or systemic corticosteroids (within 6 months of enrollment).
* Radiation proctitis or other known poorly controlled medical conditions that could interfere with bowel function.
* Patients will be excluded if using medications which are known to be affected by modest dietary changes. This will include, but is not limited to, warfarin and immunosuppressives such as cyclosporin.
* Alcohol use disorder, anorexia nervosa, autoimmune disease, bulimia, celiac disease, chronic infections, and illicit drug use.
* Major changes in dietary habits in past six months.
* Pregnancy or intent to get pregnant during study period
* Use of tobacco, including cigarettes, smokeless tobacco, cigars, and pipes within 30 days of enrollment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Change in microbiome species proportion- Oral | baseline to week 12
  Microbiome analysis will be conducted by calculating the significance in changes in the proportion of species between the groups, and by principal component analysis (PCA) to identify patterns of shift in the microbiome populations in relation to QC-induced changes.
Change in microbiome species proportion- Intestinal | baseline to week 12
  Microbiome analysis will be conducted by calculating the significance in changes in the proportion of species between the groups, and by principal component analysis (PCA) to identify patterns of shift in the microbiome populations in relation to QC-induced changes.

SECONDARY OUTCOMES:
Change in activation of the inflammasome machinery in peripheral blood cells with Pro-Il-1β | baseline to week 12
  This will be done by obtaining monocytes/macrophages from the peripheral blood and then activating them with LPS and ATP to induce up-regulation of Pro-Il-1β. Up-regulation of pro-cytokines will be performed by quantitative PCR.
Change in activation of the inflammasome machinery in peripheral blood cells with Pro-TNF-α | baseline to week 12
  This will be done by obtaining monocytes/macrophages from the peripheral blood and then activating them with LPS and ATP to induce up-regulation of Pro-TNF-α. Up-regulation of pro-cytokines will be performed by quantitative PCR.
Change in activation of the inflammasome machinery in peripheral blood cells with caspase-1 cleavage | baseline to week 12
  This will be done by obtaining monocytes/macrophages from the peripheral blood and then activating them with LPS and ATP to induce caspase-1 cleavage.
Change in activation of the inflammasome machinery in peripheral blood cells with IL-1β | baseline to week 12
  This will be done by obtaining monocytes/macrophages from the peripheral blood and then activating them with LPS and ATP to induce up-regulation of IL-1β production. Detection of cytokines will be by conventional ELISA.
Change in activation of the inflammasome machinery in peripheral blood cells with TNF-α | baseline to week 12
  This will be done by obtaining monocytes/macrophages from the peripheral blood and then activating them with LPS and ATP to induce up-regulation of TNF-α production. Detection of cytokines will be by conventional ELISA.
Change in activation of the inflammasome machinery in peripheral blood cells | baseline to week 12
  Damage associated molecular patterns (DAMPs) will be assayed.

OTHER OUTCOMES:
24-hour Dietary Recall | 2 weeks prior to baseline (at baseline)
  ASA24™ National Cancer Institute Automated Self-Administered 24-hour Dietary Recall (http://epi.grants.cancer.gov/asa24//) Questionnaire
24-hour Dietary Recall | baseline
  ASA24™ National Cancer Institute Automated Self-Administered 24-hour Dietary Recall (http://epi.grants.cancer.gov/asa24//) Questionnaire
24-hour Dietary Recall | 4 weeks
  ASA24™ National Cancer Institute Automated Self-Administered 24-hour Dietary Recall (http://epi.grants.cancer.gov/asa24//) Questionnaire
24-hour Dietary Recall | 12 weeks
  ASA24™ National Cancer Institute Automated Self-Administered 24-hour Dietary Recall (http://epi.grants.cancer.gov/asa24//) Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Shapiro, MD, Principal Investigator — Yale University; Wajahat Mehal, MD, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dioletis E, Paiva RS, Kaffe E, Secor ER, Weiss TR, Fields MR, Ouyang X, Ali A. The fermented soy beverage Q-CAN(R) plus induces beneficial changes in the oral and intestinal microbiome. BMC Nutr. 2021 Mar 4;7(1):6. doi: 10.1186/s40795-021-00408-4. PMID 33658080